CLINICAL TRIAL: NCT00303498
Title: A PHASE 2 RANDOMISED, DOUBLE-BLIND, PLACEBO-CONTROLLED EXPLORATORY EFFICACY STUDY OF SITAXSENTAN SODIUM TO IMPROVE IMPAIRED EXERCISE TOLERANCE IN SUBJECTS WITH DIASTOLIC HEART FAILURE
Brief Title: A Study of the Effectiveness of Sitaxsentan Sodium in Patients With Diastolic Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B1321006; FDHF01 (Other: Alias Study Number)
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Results first posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Diastolic Heart Failure
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitaxsentan sodium (Experimental)
  Interventions: Drug: Sitexsentin sodium
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitexsentin sodium — sitaxsentan 100 mg (target dose) 0rally once daily. A 10-week Run-In Phase was conducted where dosing commenced at 25 mg daily for 2 weeks, and then was stepped up to 50 mg daily for 2 weeks, to 75 mg daily for 2 weeks and then to 100 mg daily for 2 weeks, with an additional 2-week stabilization period (10 weeks total) to a target study dose of 100 mg daily. During the Run-In Phase, if a subject was not able to tolerate upward dose titration to the target dose of 100 mg, the investigator may have elected to continue at the current dosage or reduce the dosage of sitaxsentan or placebo to the subject's immediate prior dose. During the Maintenance Phase, subjects received the highest titrated dose reached of study drug and continued it through the last day of Week M24 of the Maintenance Phase (14 weeks)- total study drug treatment duration= 6 months
  Arms: Sitaxsentan sodium
Drug: Placebo — placebo identical to the study drug in description, dose and duration
  Arms: Placebo

SUMMARY:
The aim of this study was to determine whether long-term (≥ 6 months at the target dose) blockade of ETA receptors using sitaxsentan showed functional benefit in subjects with chronic Heart Failure and an Left Ventricular Ejection Fraction ≥50%.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older with chronic heart failure and evidence of diastolic dysfunction on echocardiogram, heart imaging, and a minimum exercise tolerance average time of 120 seconds on two treadmill tests within 2 weeks of enrollment

Exclusion Criteria:

* unstable cardiovascular disease within 4 weeks of screening, history of heart attack, cardiac by-pass surgery or percutaneous intervention, stent placement, within 3 months of screening or amyloidosis, hypertrophic obstructive or restrictive cardiomyopathy, or constrictive pericarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-03-27 (Actual); Primary Completion 2008-05-01 (Actual); Study Completion 2008-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (52):
- United States (50):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mobile Heart Specialists, PC, Mobile, Alabama
  - Preventative and Research Cardiloogy Providence Hospital, Mobile, Alabama
  - Central Arkansas Veterans HCS, Little Rock, Alaska
  - Arizona Pulmonary Specialists, LTD, Phoenix, Arizona
  - Parkview Research Center, Tucson, Arizona
  - Southwest Heart, Tucson, Arizona
  - University of Arkansas for Medical Services/Cardiology Department, Little Rock, Arkansas
  - University of Southern California Medical Center, Los Angeles, California
  - Orange County Heart Institute and Research Center, Orange, California
  - Sacramento Heart & Vascular Medical Associates, Sacramento, California
  - University of California, San Diego, California
  - Yale University School of Medicine, Cardiovascular Medicine, New Haven, Connecticut
  - Capital City Research, CCRW, Washington D.C., District of Columbia
  - Florida Heart Group Pa, Orlando, Florida
  - The University of Chicago, Chicago, Illinois
  - Methodist Medical Center, Peoria, Illinois
  - Cardiovascular Consultants of Maine, Auburn, Maine
  - Massachusetts General Hospital Pulmonary and Critical Care Unit, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - VA Med Ctr Minneapolis, Minneapolis, Minnesota
  - St. Louis University Hospital, St Louis, Missouri
  - Washington Univ. School of Medicine, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Catholic Medical Center d/b/a New England Heart Institute, Manchester, New Hampshire
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Buffalo Cardipul Assoc, Buffalo, New York
  - Columbia University Medical Center, New York Presbyterian Hospital, New York, New York
  - Capital Cardiology Associates, Troy, New York
  - Mid Carolina Cardiology, Charlotte, North Carolina
  - Mid Carolina Cardiology, Huntersville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - The Oregon Clinic, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Advanced Heart Failure & Transplant Center, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - RHJ VA Medical Center, Charleston, South Carolina
  - Black Hills Clinical Research Center, Rapid City, South Dakota
  - Stern Cardiovascular Center, Germantown, Tennessee
  - Baylor College of Medicine Pulmonary Section, Houston, Texas
  - Kelsey Seybold Clinic, Houston, Texas
  - Methodist DeBakey Heart Center, Houston, Texas
  - Intermountain Medical Center (a.k.a. LDS Hospital), Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - Fletcher Allen Health Care, Burlington, Vermont
  - Medical College of Virginia, Richmond, Virginia
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
- Canada (2):
  - St Michael's Hospital, Toronto, Ontario
  - SMBD Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Zile MR, Bourge RC, Redfield MM, Zhou D, Baicu CF, Little WC. Randomized, double-blind, placebo-controlled study of sitaxsentan to improve impaired exercise tolerance in patients with heart failure and a preserved ejection fraction. JACC Heart Fail. 2014 Apr;2(2):123-30. doi: 10.1016/j.jchf.2013.12.002. Epub 2014 Feb 26. PMID 24720918
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1321006&StudyName=A%20study%20of%20the%20effectiveness%20of%20Sitaxsentan%20Sodium%20in%20patients%20with%20Diastolic%20Heart%20Failure

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study consisted of a 10-week dose adjusting Run-In Phase followed by a 24-week Maintenance Phase.
Groups:
- Sitaxsentan: During the Run-In Phase, participants received sitaxsentan 25 milligram (mg) dose orally once daily for 2 weeks (Week 1 and Week 2). The dose was then up-titrated to 50 mg for the next 2 weeks (Week 3 and Week 4), and then to 75 mg for following 2 weeks (Week 5 and Week 6). The dose was finally up-titrated to the target study dose of 100 mg for the next 2 weeks (Week 7 and Week 8), with an additional 2-week stabilization period (up to Week 10). If a participant was unable to tolerate the upward dose titration to the target dose of 100 mg, the participant continued at the last titrated dose for the remainder of the Run-In Phase. During the Maintenance Phase, participants continued to receive the target dose of 100 mg or the maximum up-titrated Run-In Phase dose for 24 weeks.
- Placebo: Participants received placebo matched to sitaxsentan orally once daily for 34 weeks (10-Week Run-In Phase and 24-Week Maintenance Phase).
Period: Run-In-Phase (10 Weeks)
Arm/Group | Sitaxsentan | Placebo
Started | 128 | 64
Treated | 127 | 64
Completed | 104 | 56
Not Completed | 24 | 8
Not completed — Adverse Event | 5 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Sponsor Decision | 6 | 3
Not completed — Other | 4 | 1
Not completed — Treatment Interrupted More Than 7 Days | 3 | 2
Not completed — Unable to Tolerate 25 mg Dose | 1 | 0
Period: Maintenance Phase (24 Weeks)
Arm/Group | Sitaxsentan | Placebo
Started | 104 | 56
Completed | 90 | 48
Not Completed | 14 | 8
Not completed — Elevation in Liver Enzyme Values | 1 | 0
Not completed — Death | 1 | 0
Not completed — Adverse Event | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Sponsor Decision | 4 | 0
Not completed — Other | 1 | 0
Not completed — Treatment Interrupted More Than 7 Days | 1 | 2
Not completed — Required Chronic Heart Failure Treatment | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population was defined as all the participants who took at least 1 dose of study drug during the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitaxsentan | Placebo | Total
Number analyzed (Participants) | 127 | 64 | 191
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.0 (10.94) | 64.7 (9.99) | 64.9 (10.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 45 | 121
  Male | 51 | 19 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Treadmill Exercise Time at Maintenance Phase Week 24
Description: Treadmill exercise test is used to assess the functional capacity of participants with cardiac disease. Treadmill exercise test was conducted using the 2 minute incremental Naughton protocol. The Naughton protocol starts with a 2 minute warm-up. The speed of treadmill is set to 1 mile per hour (mph) and the incline is set to 0. After the warm-up, the speed is set at 2 mph for the remainder of the test. The test consists of six, 2 minute intervals. The grade starts at 0 for the first interval, and increases by 3.5 percent every 2 minutes. The change in total exercise time (in seconds) during the treadmill test was reported.
Time Frame: Baseline, Week 24 (Maintenance Phase)
Population: Intent-to-treat (ITT) population was defined as all participants who received at least 1 dose of study drug and had at least 1 valid treadmill test value at baseline and post-baseline during maintenance phase. Last observation carried forward (LOCF) method was used to impute missing values.
Measure: Median (Full Range); unit: Seconds
Arm/Group | Sitaxsentan | Placebo
Number analyzed (Participants) | 96 | 52
Seconds
  Baseline | 424.5 [121 to 706] | 485.0 [126 to 693]
  Change at Week 24 | 89.5 [-235 to 549] | 37.0 [-141 to 490]
Statistical Analysis 1: Comparison: Sitaxsentan vs Placebo; The median of the treatment difference was calculated using the Hodges-Lehmann estimator; Test type: Superiority or Other; p = 0.0302, ANCOVA; Change at Week 24: P-value was obtained from the non-parametric analysis of covariance (ANCOVA) controlling for baseline treadmill exercise time; Median Difference (Net) = 43.0

2. Secondary Outcome: Change From Baseline in Ratio of Transmitral Inflow Velocity (E) to Early Diastolic Velocity of the Mitral Annulus (E') at Maintenance Phase Week 24
Description: Ratio of E to E' is used as a predictor of first cardiac events. Ratio of E to E' was measured using imaging techniques based on Doppler principles. Transmitral inflow velocity was measured by Doppler echocardiography (ECHO) and the early diastolic velocity of the mitral annulus was measured by tissue Doppler imaging (TDI).
Time Frame: Baseline, Week 24 (Maintenance Phase)
Population: ITT population was defined as all the participants who received at least 1 dose of study drug and had at least 1 valid treadmill test value at baseline and post-baseline during maintenance phase. Here, "Overall Number of Participants Analyzed" signifies number of participants who were evaluable for this outcome measure and 'Number Analyzed' signifies the participants who were evaluable at the specified time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Sitaxsentan | Placebo
Number analyzed (Participants) | 73 | 49
Ratio
  Baseline | 13.72 (6.975) | 14.45 (6.565)
  Change at Week 24: number analyzed (Participants) | 55 | 37
  Change at Week 24 | -0.12 (4.404) | 0.38 (4.498)
Statistical Analysis 1: Comparison: Sitaxsentan vs Placebo; Test type: Superiority or Other; p = 0.4950, ANCOVA; Change at Week 24: P-value was calculated from an ANCOVA with effect for treatment and baseline value as a covariate; Mean Difference (Net) = -0.5

3. Secondary Outcome: Change From Baseline in Left Ventricular Mass at Maintenance Phase Week 24
Description: Left ventricular mass was used as a parameter for the assessment of cardiac function. An increase in left ventricular mass leads to ventricular hypertrophy which is a prognostic factor of cardiovascular morbidity and mortality. Left ventricular mass was measured by ECHO, which was calculated as (1.04 * [{left ventricular end diastolic diameter (LVEDD) + septal diastolic thickness + post wall diastolic thickness}^3 - LVEDD^3]) * 0.8 + 0.6. Left ventricular mass was assessed for the two ECHO modes: parasternal long-axis two dimensional (PLAX 2D) mode and parasternal short-axis view motion (PSAX M) mode.
Time Frame: Baseline, Week 24 (Maintenance Phase)
Population: ITT population defined as all participants who received at least 1 dose of study drug and had at least 1 valid treadmill test value at baseline and post-baseline during maintenance phase. Here, "Overall Number of Participants Analyzed" signifies number of participants who were evaluable for this outcome measure and 'Number Analyzed' signifies the participants who were evaluable at the specified time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: Centimeter^3
Arm/Group | Sitaxsentan | Placebo
Number analyzed (Participants) | 55 | 31
Centimeter^3
  Baseline: PLAX 2D mode | 217.73 (80.467) | 226.14 (83.415)
  Baseline: PSAX M-mod: number analyzed (Participants) | 26 | 19
  Baseline: PSAX M-mod | 229.88 (70.251) | 229.19 (108.891)
  Change at Week 24: PLAX 2D mode: number analyzed (Participants) | 35 | 19
  Change at Week 24: PLAX 2D mode | 3.09 (43.647) | -7.52 (42.582)
  Change at Week 24: PSAX M-mode: number analyzed (Participants) | 9 | 6
  Change at Week 24: PSAX M-mode | 5.60 (45.641) | 4.83 (10.565)
Statistical Analysis 1: Comparison: Sitaxsentan vs Placebo; Change at Week 24 for PLAX 2D mode; Test type: Superiority or Other; p = 0.3874, ANCOVA; P-value was calculated from an ANCOVA with effect for treatment and baseline value as a covariate; Mean Difference (Net) = 10.6
Statistical Analysis 2: Comparison: Sitaxsentan vs Placebo; Change at Week 24 for PSAX M-mode; Test type: Superiority or Other; p = 0.7038, ANCOVA; P-value was calculated from an ANCOVA with effect for treatment and baseline value as a covariate; Mean Difference (Net) = 0.8

4. Secondary Outcome: Change From Baseline in Minnesota Living With Heart Failure (MLHF) Questionnaire - Quality of Life (QoL) Total Score at Maintenance Phase Week 24
Description: The MLHF is a 21-item questionnaire which used to evaluate QoL in participants suffering from heart failure. The participants were asked to evaluate how their heart condition affected their life during the past month. Each of the 21 items were assessed on a 6-point scale, where 0 = no affect and 5 = very much affected. The MLHF QoL total score was calculated as the sum of the 21 individual QoL questions. The MLHF QoL total score ranged from 0 to 105, where higher scores indicated worse health condition.
Time Frame: Baseline, Week 24 (Maintenance Phase)
Population: ITT population. Here, "Overall Number of Participants Analyzed" signifies number of participants who were evaluable for this outcome measure. LOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sitaxsentan | Placebo
Number analyzed (Participants) | 91 | 51
Units on a scale
  Baseline | 43.79 (26.100) | 37.67 (23.559)
  Change at Week 24 | -8.20 (21.493) | -6.31 (18.909)
Statistical Analysis 1: Comparison: Sitaxsentan vs Placebo; Test type: Superiority or Other; p = 0.8998, ANCOVA; P-value was calculated from an ANCOVA with effect for treatment and baseline value as a covariate; Mean Difference (Net) = -1.9

5. Secondary Outcome: Change From Baseline in Minnesota Living With Heart Failure (MLHF) Questionnaire - Quality of Life (QoL) Physical Score at Maintenance Phase Week 24
Description: The MLHF is a 21-item questionnaire which is used to evaluate QoL in participants suffering from heart failure. The participants were asked to evaluate how their heart condition affected their life during the past month. Each of the 21 items were assessed on a 6-point scale, where 0 = no affect and 5 = very much affected. The MLHF QoL physical score was calculated as the sum of the 8 physical domain QoL questions. The MLHF QoL physical score ranged from 0 to 40, where higher scores indicated worse health condition.
Time Frame: Baseline, Week 24 (Maintenance Phase)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sitaxsentan | Placebo
Number analyzed (Participants) | 94 | 52
Units on a scale
  Baseline | 21.73 (11.740) | 18.85 (10.151)
  Change at Week 24 | -4.06 (10.365) | -2.35 (8.753)
Statistical Analysis 1: Comparison: Sitaxsentan vs Placebo; Test type: Superiority or Other; p = 0.7245, ANCOVA; P-value was calculated from an ANCOVA with effect for treatment and baseline value as a covariate; Mean Difference (Net) = -1.7

6. Secondary Outcome: Change From Baseline in Minnesota Living With Heart Failure (MLHF) Questionnaire - Quality of Life (QoL) Emotional Score at Maintenance Phase Week 24
Description: The MLHF is a 21-item questionnaire which is used to evaluate QoL in participants suffering from heart failure. The participants were asked to evaluate how their heart condition affected their life during the past month. Each of the 21 items were assessed on a 6-point scale, where 0 = no affect and 5 = very much affected. The MLHF QoL emotional score was calculated as the sum of the 5 emotional domain QoL questions. The MLHF QoL emotional score ranged from 0 to 25, where higher scores indicated worse health condition.
Time Frame: Baseline, Week M24 (Maintenance Phase)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sitaxsentan | Placebo
Number analyzed (Participants) | 93 | 52
Units on a scale
  Baseline | 8.97 (7.562) | 7.37 (6.914)
  Change at Week 24 | -1.87 (6.094) | -1.40 (5.815)
Statistical Analysis 1: Comparison: Sitaxsentan vs Placebo; Test type: Superiority or Other; p = 0.8649, ANCOVA; P-value was calculated from an ANCOVA with effect for treatment and baseline value as a covariate; Mean Difference (Net) = -0.5

7. Secondary Outcome: Number of Participants With Change From Baseline in New York Heart Association (NYHA) Functional Class at Maintenance Phase Week 24
Description: Participants were classified by NYHA functional class. NYHA class I: participants with cardiac disease but without resulting limitations of physical activity, NYHA class II: participants with cardiac disease resulting in slight limitation of physical activity, NYHA class III: participants with cardiac disease resulting in marked limitation of physical activity, NYHA class IV: participants with cardiac disease resulting in inability to carry on any physical activity without discomfort. Baseline was reported by NYHA functional class and the change from baseline in the functional class was reported as improvement (positive change from baseline), no change and deterioration (negative change from baseline).
Time Frame: Baseline, Week 24 (Maintenance Phase)
Population: ITT population. LOCF method was used to impute missing values.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitaxsentan | Placebo
Number analyzed (Participants) | 96 | 52
Participants
  Baseline: Class II | 58 | 27
  Baseline: Class III | 38 | 25
  Improvement | 30 | 18
  No change | 60 | 34
  Deterioration | 6 | 0
Statistical Analysis 1: Comparison: Sitaxsentan vs Placebo; Change at Week 24; Test type: Superiority or Other; p = 0.5909, Cochran-Mantel-Haenszel — The statistical analysis (P value) was performed on the composite change for all categories

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sitaxsentan | Placebo
Serious Adverse Events (participants affected / at risk) | 25/127 | 16/64
Other Adverse Events (participants affected / at risk) | 107/127 | 54/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitaxsentan (N=127) | Placebo (N=64)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 2
Coronary artery disease (Cardiac disorders) | 3 | 0
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 3 | 2
Generalised oedema (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Incision site infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1
Sepsis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Bladder disorder (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Colpocele (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal hernia repair (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitaxsentan (N=127) | Placebo (N=64)
Anaemia (Blood and lymphatic system disorders) | 7 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 3 | 3
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bundle branch block right (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Cardiac flutter (Cardiac disorders) | 2 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Cyanosis (Cardiac disorders) | 1 | 0
Low cardiac output syndrome (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 6 | 8
Pulmonary valve disease (Cardiac disorders) | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Ear pain (Ear and labyrinth disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Thyroid cyst (Endocrine disorders) | 1 | 0
Blindness transient (Eye disorders) | 0 | 1
Eye allergy (Eye disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Posterior capsule rupture (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal hernia (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 2 | 5
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 4
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 10 | 4
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 5 | 3
Adverse drug reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Chest discomfort (General disorders) | 4 | 1
Chest pain (General disorders) | 7 | 4
Chills (General disorders) | 2 | 1
Fatigue (General disorders) | 10 | 4
Ill-defined disorder (General disorders) | 0 | 1
Malaise (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 3 | 2
Oedema (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 20 | 8
Pain (General disorders) | 3 | 0
Peripheral swelling (General disorders) | 3 | 2
Pyrexia (General disorders) | 1 | 1
Swelling (General disorders) | 0 | 1
Thirst (General disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 2
Acarodermatitis (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 3 | 1
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 1
Ear infection (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 1 | 2
Fungal skin infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 3 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 4 | 2
Kidney infection (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 2
Nail infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 6 | 4
Oral herpes (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 5 | 2
Tooth abscess (Infections and infestations) | 2 | 0
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 13 | 3
Urinary tract infection (Infections and infestations) | 12 | 5
Wound infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 2
Eschar (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 3 | 2
Blood glucose abnormal (Investigations) | 0 | 1
Blood glucose fluctuation (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 1 | 1
Blood potassium increased (Investigations) | 1 | 1
Blood pressure increased (Investigations) | 1 | 0
Blood pressure orthostatic increased (Investigations) | 1 | 0
Clostridium test (Investigations) | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 1 | 0
Eosinophil count increased (Investigations) | 3 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 1
Haematocrit decreased (Investigations) | 2 | 1
Haemoglobin decreased (Investigations) | 3 | 2
Heart rate decreased (Investigations) | 1 | 0
Heart rate increased (Investigations) | 0 | 1
Helicobacter test positive (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 2 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Occult blood positive (Investigations) | 0 | 2
Pedal pulse decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Red cell distribution width increased (Investigations) | 0 | 1
Renal function test abnormal (Investigations) | 0 | 1
Reticulocyte count increased (Investigations) | 0 | 1
Weight increased (Investigations) | 1 | 4
White blood cell count increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 4 | 1
Gout (Metabolism and nutrition disorders) | 2 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 4
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 5
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 4
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Eyelid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 10 | 6
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 9 | 11
Hypoaesthesia (Nervous system disorders) | 2 | 1
Lethargy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 2 | 2
Poor quality sleep (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 2 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 2 | 1
Somnolence (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 2 | 3
Tremor (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 3
Depression (Psychiatric disorders) | 0 | 2
Dissociative fugue (Psychiatric disorders) | 1 | 0
Euphoric mood (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 4
Nightmare (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 2
Renal failure (Renal and urinary disorders) | 2 | 0
Urine odour abnormal (Renal and urinary disorders) | 1 | 0
Breast enlargement (Reproductive system and breast disorders) | 0 | 1
Breast haemorrhage (Reproductive system and breast disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 2 | 0
Breast tenderness (Reproductive system and breast disorders) | 1 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 4
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Cataract operation (Surgical and medical procedures) | 1 | 0
Lung operation (Surgical and medical procedures) | 0 | 1
Oral surgery (Surgical and medical procedures) | 0 | 1
Sinus operation (Surgical and medical procedures) | 1 | 0
Synovectomy (Surgical and medical procedures) | 1 | 0
Toe operation (Surgical and medical procedures) | 0 | 1
Uterine dilation and curettage (Surgical and medical procedures) | 0 | 1
Flushing (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 3
Hypertension (Vascular disorders) | 4 | 3
Hypotension (Vascular disorders) | 8 | 2
Lymphoedema (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.